CLINICAL TRIAL: NCT04595955
Title: Effectiveness of the Digital Patient Platform CMyLife for Patients With Chronic Myeloid Leukemia
Brief Title: Effects of a Digital Patient Platform (CMyLife) for Patients With Chronic Myeloid Leukemia (CML) on Information Provision, Patient Empowerment, Medication Compliance, Guideline Adherence and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: RU_23-08-20_LV
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Neoplasms; Chronic Myeloid Leukemia; Patient Portals; Telemedicine
MeSH Terms: conditions — Neoplasms; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This arm uses the CMyLife platform for at least 6 months
  Interventions: Other: CMyLife
- Control group (No Intervention): This arm does not use the CMyLife platform

INTERVENTIONS:
Other: CMyLife — CMyLife is a digital patient platform for Patients With Chronic Myeloid Leukemia.
  Arms: Intervention group

SUMMARY:
A controlled before-after study is performed in order to gain insights into the effectiveness of the CMyLife platform in terms of medication compliance, guideline adherence, quality of life, information provision and patient empowerment. Participants who agreed to use the CMyLife platform for at least 6 months, were enrolled in the treatment group and participants who did not agree to use the platform were enrolled in the control group. After signing informed consent, participants received a baseline questionnaire by mail. Upon completion of the baseline questionnaire, participants used (intervention group) or did not use (control group) the CMyLife platform for at least 6 months, after which they were asked to complete the post-intervention questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed CML patients in chronic phase CML
* Participants were treated with first or second line TKI's at the haematology department of the participating hospitals. Patients treated with second line TKI's were only allowed to participate if they switched TKI's as a result of side effects and not if they did not respond to the first line TKI

Exclusion Criteria:

* Participants in acceleration phase
* Participants in blastcrise
* Participants with planned pregnancy in the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
the information received by CML patients | at baseline
  To evaluate the information received by participants the EORTC QLQ-INFO25 was used
the information received by CML patients | 6 months after baseline
  To evaluate the information received by participants the EORTC QLQ-INFO25 was used
patient empowerment | at baseline
  The Patient Activation Measure was used to gain more insight into how and to what extent the participant believed that he/she is able to improve his/her own health
patient empowerment | 6 months after baseline
  The Patient Activation Measure was used to gain more insight into how and to what extent the participant believed that he/she is able to improve his/her own health
eHealth Literacy | at baseline
  Participants' ability to find and evaluate online health information was measured using the eHealth Literacy Scale
eHealth Literacy | 6 months after baseline
  Participants' ability to find and evaluate online health information was measured using the eHealth Literacy Scale
medication compliance | at baseline
  medication compliance of participants was measured using the Medication Adherence Rating Scale
medication compliance | 6 months after baseline
  medication compliance of participants was measured using the Medication Adherence Rating Scale
guideline adherence | at baseline
  guideline adherence was measured using the frequency of BCR-ABL1 value checks
guideline adherence | 6 months after baseline
  guideline adherence was measured using the frequency of BCR-ABL1 value checks
Patients' experiences | at baseline
  Participants' experiences with the care and information they receive in hospitals for their CML were measured using Patient Reported Experience Measures
Patients' experiences | 6 months after baseline
  Participants' experiences with the care and information they receive in hospitals for their CML were measured using Patient Reported Experience Measures
Quality of life of CML patients: EORTC QLQ-C30 | at baseline
  Quality of life of participants was measured using the EORTC QLQ-C30
Quality of life of CML patients: EORTC QLQ-C30 | 6 months after baseline
  Quality of life of participants was measured using the EORTC QLQ-C30
disease (CML) specific quality of life: EORTC QLQ-CML24 | at baseline
  disease specific quality of life of participants was measured using the EORTC QLQ-CML24
disease (CML) specific quality of life: EORTC QLQ-CML24 | 6 months after baseline
  disease specific quality of life of participants was measured using the EORTC QLQ-CML24

SECONDARY OUTCOMES:
Familiarity with CML related concept: Philadelphia chromosome | at baseline
  % of participants who are not (at all) familiar with the concept Philadelphia chromosome
Familiarity with CML related concept: Philadelphia chromosome | 6 months after baseline
  % of participants who are not (at all) familiar with the concept Philadelphia chromosome
Familiarity with CML related concept: BCR-ABL | at baseline
  % of participants who are not (at all) familiar with the concept BCR-ABL
Familiarity with CML related concept: BCR-ABL | 6 months after baseline
  % of participants who are not (at all) familiar with the concept BCR-ABL
Familiarity with CML related concept: tyrosine kinase inhibitor | at baseline
  % of participants who are not (at all) familiar with the concept tyrosine kinase inhibitor
Familiarity with CML related concept: tyrosine kinase inhibitor | 6 months after baseline
  % of participants who are not (at all) familiar with the concept tyrosine kinase inhibitor
Familiarity with CML related concept: remission | at baseline
  % of participants who are not (at all) familiar with the concept remission
Familiarity with CML related concept: remission | 6 months after baseline
  % of participants who are not (at all) familiar with the concept remission
Familiarity with CML related concept: log reduction | at baseline
  % of participants who are not (at all) familiar with the concept log reduction
Familiarity with CML related concept: log reduction | 6 months after baseline
  % of participants who are not (at all) familiar with the concept log reduction
Familiarity with CML related concept: hematologic response/remission | at baseline
  % of participants who are not (at all) familiar with the concept hematologic response/remission
Familiarity with CML related concept: hematologic response/remission | 6 months after baseline
  % of participants who are not (at all) familiar with the concept hematologic response/remission
Familiarity with CML related concept: cytogenetic response/remission | at baseline
  % of participants who are not (at all) familiar with the concept cytogenetic response/remission
Familiarity with CML related concept: cytogenetic response/remission | 6 months after baseline
  % of participants who are not (at all) familiar with the concept cytogenetic response/remission
Familiarity with CML related concept: molecular response/remission | at baseline
  % of participants who are not (at all) familiar with the concept molecular response/remission
Familiarity with CML related concept: molecular response/remission | 6 months after baseline
  % of participants who are not (at all) familiar with the concept molecular response/remission
Familiarity with CML related concept: major molecular remission | at baseline
  % of participants who are not (at all) familiar with the concept major molecular remission
Familiarity with CML related concept: major molecular remission | 6 months after baseline
  % of participants who are not (at all) familiar with the concept major molecular remission
Familiarity with CML related concept: complete cytogenetic remission | at baseline
  % of participants who are not (at all) familiar with the concept complete cytogenetic remission
Familiarity with CML related concept: complete cytogenetic remission | 6 months after baseline
  % of participants who are not (at all) familiar with the concept complete cytogenetic remission
Familiarity with CML related concept: treatment free remission | at baseline
  % of participants who are not (at all) familiar with the concept treatment free remission
Familiarity with CML related concept: treatment free remission | 6 months after baseline
  % of participants who are not (at all) familiar with the concept treatment free remission
Familiarity with CML related concept: Hematon | at baseline
  % of participants who are not (at all) familiar with the concept hematon
Familiarity with CML related concept: Hematon | 6 months after baseline
  % of participants who are not (at all) familiar with the concept hematon

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
The plan is to share IPD when Radboudumc arranged this possibility.

REFERENCES:
- [Derived] Verweij L, Ector GICG, Smit Y, van Vlijmen B, van der Reijden BA, Hermens RPMG, Blijlevens NMA. Effectiveness of digital care platform CMyLife for patients with chronic myeloid leukemia: results of a patient-preference trial. BMC Health Serv Res. 2023 Mar 8;23(1):228. doi: 10.1186/s12913-023-09153-9. PMID 36890512